CLINICAL TRIAL: NCT03246048
Title: Predicting Outcomes in Hepatitis C Patients With Compensated Advanced Chronic Liver Disease Cured With New Antivirals
Brief Title: Long Term Follow-up of Hepatitis C Cured Patients
Status: Completed | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PR(AG)136/2017
Record Dates: First submitted 2017-08-08; First posted 2017-08-11 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Chronic Hepatitis C; Chronic Liver Disease; Cirrhosis
MeSH Terms: conditions — Hepatitis C, Chronic; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Objectives:

The general objective of the present project is to gain a better understanding of disease outcome in cACLD patients treated with the new oral DAA. In particular, the project will focus on:

- To evaluate the long term prognosis of patients with compensated advanced chronic liver disease (cACLD) who achieve sustained virological response (SVR) after the new oral direct-acting antiviral agents (DAA), and determine clinical and elastographic basal and follow-up parameters to identify low and high risk groups of developing liver-related decompensation.

Methods:

Prospective cohort study in patients with cACLD in whom basal and annual clinical features and liver stiffness measurements (LSM) will be performed, and survival free of liver-related events will be analyzed.

DETAILED DESCRIPTION:
HYPOTHESIS:

- The prognosis of cACLD patients who achieve SVR will improve during follow-up and this will be reflected in an improvement in liver and spleen stiffness and reduction of liver-related events. However, on an individual basis, because of many confounding factors, predictability is unknown.

OBJECTIVES:

The general objective of the present project is to gain a better understanding of disease outcome in cACLD patients treated with the new oral DAA. In particular, the project will focus on to determine simple clinical and elastographic basal and follow-up parameters to identify low and high risk groups for developing liver-related decompensation in cACLD patients who achieve SVR after DAA therapy. As a consequence of this, to provide guidance to clinicians to decide which cACLD patients should be indefinitely followed and which ones can be discharged from follow up, and also provide solid information to patients regarding the possible outcome of their cACLD after SVR.

* Study design: Prospective cohort study in an academic center to evaluate long term prognosis of patients with cACLD who achieve SVR after DAA therapy.
* Research subjects: All consecutive patients meeting inclusion criteria who have received DAA therapy from 1st January 2015 to 31st March 2016.
* Variables: Variables will be collected at baseline and annually for a period of 5 years. Basal data on genotype/subtype, interleukin 28B, viremia, type and duration of therapy. Data of liver function (INR, albumin, bilirubin), platelet count, aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (AP), gamma-glutamyltransferase (GGT), US findings (spleen size, collaterals), liver and spleen stiffness, body mass index (BMI), presence of metabolic syndrome factors (diabetes, dyslipemia, hypertension), alcohol and tabacco use, treatment with statins and development of liver-related events. The subgroup of patients with known esophageal varices prior to therapy will receive a second endoscopy 12-18 months after finishing therapy. Liver biopsies will be performed (after consent) at the end of follow-up (5 years) in the group of patients who will be candidates for being discharged (LSM<10 kPa) to ensure cirrhosis regression and learn about the correlation between LSM and histology after SVR.
* Data collection methods and analysis: Patients will be monitored at the outpatient clinics every 6 months as per usual clinical practice. Every 6 months, clinical data, laboratory tests and abdominal US will be obtained. Liver and spleen stiffness (Fibroscan, Echosens) will be performed annually after finishing treatment by an experienced member (MP), using usual quality criteria. Spleen stiffness measurements will be performed under US spleen localization and with the same device and conditions than liver stiffness. All data will be registered in a database.

ELIGIBILITY:
Inclusion Criteria:

1. Patients having suggestive or highly suggestive cACLD defined as LSM 10-15 kPa or LSM ≥15 kPa, respectively. Patients with suggestive cACLD (LSM 10-15 kPa) will be divided in two subgroups depending on the presence of at least one of the following: gastroesophageal varices, hepatic venous pressure gradient (HVPG) >5 mmHg, nodular liver or collateral circulation in US, splenomegaly (>=13 cm) or platelet count <150,000. Patients with suggestive cACLD (LSM 10-15 kPa) and none of the prior characteristics will form the subgroup of occult cACLD.
2. Age between 18-85 years old.
3. SVR after antiviral therapy.
4. Signed informed consent.

Exclusion Criteria:

1. History of liver decompensation.
2. Hepatitis B virus coinfection.
3. HIV infection.
4. Prior liver transplantation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients meeting inclusion criteria who have received DAA therapy from 1st January 2015 to 31st March 2016.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Incidence of liver decompensation and/or death and hepatocellular carcinoma | 5 years
  Incidence of liver related events (decompensation and hepatocellular carcinoma) during follow-up

SECONDARY OUTCOMES:
Correlate values of liver stiffness with histology changes at the end of follow up | 5 years
  Correlate liver fibrosis in liver biopsy with liver stiffness cut-offs.

CONTACTS AND LOCATIONS:
Overall Officials: Joan Genescà, Principal Investigator — Hospital Vall d'Hebron